CLINICAL TRIAL: NCT02723240
Title: A Two-part, Phase I Open Label, Dose Escalation and Expansion Study to Assess Safety, Pharmacokinetics and Clinical Activity of NUC-3373, a Nucleotide Analogue, in Participants With Advanced Solid Tumours
Brief Title: NUC-3373 in Advanced Solid Tumours
Acronym: NuTide:301
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_074; 2015-002250-13 (EudraCT Number)
Record Dates: First submitted 2015-12-08; First posted 2016-03-30 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2021-04

CONDITIONS: Cancer
Keywords: NUC-3373; Dose escalation; Nucleotide Analogue
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Part 1 (weekly administration) NUC-3373 125mg/m2 (Experimental): NUC-3373 125mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 250mg/m2 (Experimental): NUC-3373 250mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 500mg/m2 (Experimental): NUC-3373 500mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 750mg/m2 (Experimental): NUC-3373 750mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 1125mg/m2 (Experimental): NUC-3373 1125mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 1500mg/m2 (Experimental): NUC-3373 1500mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 1875mg/m2 (Experimental): NUC-3373 1875mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 2500mg/m2 (Experimental): NUC-3373 2500mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 1 (weekly administration) NUC-3373 3250mg/m2 (Experimental): NUC-3373 3250mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 8, Day 15, Day 22 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 2 (two weekly administration) NUC-3373 1500mg/m2 (Experimental): NUC-3373 1500mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 15 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 2 (two weekly administration) NUC-3373 1875mg/m2 (Experimental): NUC-3373 1875mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 15 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373
- Part 2 (two weekly administration) NUC-3373 2500mg/m2 (Experimental): NUC-3373 2500mg/m2 solution for injection/infusion IV Infusion on Day 1, Day 15 (28 day cycle).
  Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.
  Interventions: Drug: NUC-3373

INTERVENTIONS:
Drug: NUC-3373

SUMMARY:
A two-part, phase I open label, dose escalation and expansion study to assess safety, pharmacokinetics and clinical activity of NUC-3373, a nucleotide analogue, in participants with advanced solid tumours.

DETAILED DESCRIPTION:
This is a two-part, Phase I dose escalation study of NUC-3373 (a pyrimidine nucleotide analogue) as a single agent, administered weekly or fortnightly as an I.V. (intravenous) infusion.

In both parts participants will undergo evaluations of the safety, PK (pharmacokinetics), PD (pharmacodynamics) and anti-tumour efficacy of NUC-3373

• Participants may continue to receive NUC-3373 until disease progression or unacceptable toxicity occurs.

Part 1: Establish the RP2D (recommended phase two dose) and assess the safety and tolerability for single agent NUC-3373 administered as an I.V. infusion on day 1, 8, 15, 22 of a 28-day cycle. Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs. The RP2D will be determined by dose escalation with sequential participants receiving increasing doses of NUC-3373 in a standard '3 + 3' cohort design.

Part 2: Establish the RP2D and assess the safety and tolerability for single agent NUC-3373 administered as a fortnightly I.V. infusion on day 1 and 15 of a 28-day cycle. Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs. The RP2D will be determined by dose escalation with sequential participants receiving increasing doses of NUC-3373 in a standard '3 + 3' cohort design.

Finally, to assess preliminary efficacy signals and further characterise the safety profile, expansion cohorts of up to 20 additional participants per cohort will receive the RP2D of NUC-3373 as determined in Part 1 and Part 2 of the study. Participants can remain on study and receive treatment until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Diagnosis: Histologically confirmed diagnosis of solid tumour, which is not amenable to standard chemotherapy, is refractory to standard chemotherapy or for which no standard chemotherapy exists.
3. Age ≥ 18 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
5. Life expectancy of ≥ 12 weeks.
6. Participants must have measurable disease per RECIST criteria and/or evaluable disease (evaluable: cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions which do not fulfil RECIST criteria for measurable disease).
7. Adequate bone marrow function as defined by: WBC of ≥ 3 x109/L, ANC of ≥ 1.5 x 109/L, platelet count of ≥ 100 x 109/L, and haemoglobin of ≥ 9g/dL.
8. Adequate liver function, as determined by: Serum total bilirubin ≤1.5 x ULN, AST and ALT ≤ 2.5 x ULN.
9. Adequate renal function as defined by serum creatinine within ≤ 1.5 x ULN upper limits of normal or calculated clearance ≥50 ml/min/1.73 m2. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (using the Cockcroft-Gault formula). For subjects with a Body Mass Index (BMI) >30 kg/m2, lean body weight should be used instead
10. Left Ventricular Ejection Fraction (LVEF) ≥50% on echocardiogram
11. Ability to comply with protocol requirements.
12. Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the first scheduled IMP administration at Cycle 1 Day 1. .

Exclusion Criteria:

1. History of allergic reactions attributed to previous 5-FU or capecitabine treatment.
2. History of allergic reactions to any of the components of the diluent solutions supplied with NUC-3373.
3. Symptomatic CNS or leptomeningeal metastases.
4. Participants with a history of myocardial infarction within the last 5 years or with significant cardiac arrhythmias requiring medication or pacemaker.
5. Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy for bone pain), immunotherapy or any other anticancer agent within 28 days of first administration of the IMP.

   * For nitrosoureas and mitomycin C within 6 weeks of first administration of IMP.
   * For hormone or biological therapy within 14 days of first administration of IMP.
6. Prior toxicities from chemotherapy or radiotherapy which have not regressed to Grade ≤ 1 severity (NCI-CTCAE version 4.0) apart from renal function (provided inclusion criteria 9 is met), neuropathy and alopecia.
7. Another active cancer excluding basal cell carcinoma or intraepithelial neoplasia (CIN/cervical in situ or melanoma in situ).
8. Participants with uncontrolled concomitant illness, active infection requiring i.v. antibiotics, or uncontrolled infections, or a fever >38.5°C on the day of scheduled dosing.
9. Participants with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the CI or delegates opinion would be likely to interfere with a participant's participation in the study, or with the interpretation of the results.
10. Known HIV or known active Hepatitis B or C.
11. Any condition (e.g. known or suspected poor compliance, psychological instability, geographical location, etc.) that, in the judgment of the CI or delegates may affect the participant's ability to sign the informed consent and undergo study procedures.
12. All men or women of reproductive potential, unless using at least two contraceptive precautions, one of which must be from the list below, the other must be a condom*1 or abstaining from sexual intercourse, until six months after treatment has ended:

    * Combined (oestrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation: either oral, intravaginal or transdermal.
    * Progesterone-only hormonal contraception associated with inhibition of ovulation: either oral, injectable or implantable.
    * Intra-uterine device (IUD)
    * Intra-uterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomised partner*2
    * Sexual abstinence*3
13. Participants who are currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-01; Primary Completion 2020-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
To establish the recommended Phase 2 Dose (RP2D) of NUC-3373 that will optimise the risk/benefit reward for the participants, administered weekly (Part 1) and when administered fortnightly (Part 2), as a single I.V. infusion. | To decide if the next cohort can be opened at a higher dose level, the Trial Management Group (TMG) will review available data (e.g. safety profile) once all participants in the preceding cohort have completed the first cycle through to Day 28.
  The RP2D is the most appropriate dose that will optimise the risk/benefit reward for the participants. RP2D determination will take into consideration the plasma PK, PD assessments, the nature of the PK/PD relationship, any efficacy signals or any adverse events observed during the conduct of the dose-escalation and the available non clinical data.
  The RP2D will be determined by dose escalation with sequential participants receiving increasing doses of NUC-3373 in a standard '3 + 3' cohort design. Dose escalation will stop when the Maximum Tolerated Dose (MTD)/RP2D have been defined for that Part or a decision is made by the Trial Management Group to halt enrolment.

SECONDARY OUTCOMES:
Dose Limiting Toxicities (DLT) to assess the tolerability of NUC-3373 | Assessment starts at first IMP administration (Cycle 1 Day 1) until the first cycle completion (Day 28)
  A DLT is defined, following case causality assessment of 'Definite', 'Probable', or 'Possible' and as such may be related to the IMP:
  * Greater than or equal to Grade 3 non-haematological toxicity (e.g. mucositis, stomatitis and hand-foot syndrome) (excluding nausea/vomiting/diarrhoea or rash that responds to standard medical treatment or as allowed by eligibility criteria e.g. elevated LFTs in participants with liver metastases).
  * Greater than or equal to Grade 3 nausea/vomiting/diarrhoea or rash that occurs despite standard medical treatment for such AEs (see 3.6.1).
  * Grade 4 neutropaenia.
  * Febrile neutropaenia.
  * Grade 4 thrombocytopaenia.
  * Inability to begin next dose of treatment within 14 days of the scheduled dosing due to unresolved toxicity related to NUC-3373.
  * Either isolated or recurrent (i.e., cardiac, renal, neurologic) toxicity that is judged by the CI and/or TMG to be a DLT.
Dose Limiting Toxicities (DLT) and SAEs/AEs to assess the safety of NUC-3373 | Adverse event monitoring starts at IMP administration (Day 1) until 28 days after the final dose of IMP has been administered.
  All adverse events (AEs) using NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) v4.0 will be listed and summarised by descriptive statistics for all patients grouped by each dose level for each part. During treatment participants will be reviewed on a weekly basis during the first cycle and on the day of treatment. Additional visits may be arranged at the investigator's discretion. The categories will be AE, AE with CTCAE grade >3 and serious adverse events (SAE) related or not related to NUC-3373. Data presented throughout study completion, SAEs reviewed in real-time, TMG review all data (monthly meeting on average).
Analysis of NUC-3373 metabolites in plasma to determine Area under the curve (AUC) | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  To determine the pharmacokinetics (PK) of NUC-3373 and key metabolites, samples taken:
  * Part 1: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in plasma to determine Peak Plasma Concentration (Cmax) | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  To determine the pharmacokinetics (PK) of NUC-3373 and key metabolites, samples taken:
  * Part 1: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in plasma to determine Clearance | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  To determine the pharmacokinetics (PK) of NUC-3373 and key metabolites, samples taken:
  * Part 1: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then samples taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in plasma to determine plasma half T1/2 | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  Analysis of NUC-3373 metabolites in PBMC, to determine the pharmacokinetics (PK) of NUC-3373 and key metabolites. Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in PBMC to determine Peak Plasma Concentration (Cmax) | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  Analysis of NUC-3373 metabolites in PBMC, to determine the pharmacokinetics (PK) of NUC-3373 and key metabolites. Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in PBMC to determine Area under the curve (AUC) | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  Analysis of NUC-3373 metabolites in PBMC, to determine the pharmacokinetics (PK) of NUC-3373 and key metabolites.
  Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in PBMC determine plasma half T1/2 | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  Analysis of NUC-3373 metabolites in PBMC, to determine the pharmacokinetics (PK) of NUC-3373 and key metabolites.
  Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Analysis of NUC-3373 metabolites in PBMC to determine Clearance | PK samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  Analysis of NUC-3373 metabolites in PBMC, to determine the pharmacokinetics (PK) of NUC-3373 and key metabolites.
  Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
    * Urine samples taken: 0-6 and 6-24 hour urine collection starting from beginning of IMP infusion.
Measuring the ratio between the intracellular dTMP and dUMP concentrations. | PD samples will be collected on Cycle 1 Day 1 and Cycle 1 Day 15
  For analysis on the effect of NUC-3373 on thymidylate synthetase activity in the PBMC to determine the pharmacodynamics (PD) of NUC-3373. We will use a sensitive and specific liquid chromatography-mass spectrometry method for quantification of these intracellular metabolites.
  The unmodified TS (TS-U) and the TS in ternary complexes (TS-T) will be assessed using Western Blotting approach.
  Samples taken:
  * Part 1: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
  * Part 2: Pre-dose sample; Then sample taken immediately after the drug has cleared the infusion line; then at 5 minutes; 15 minutes; 30 minutes; 45 minutes, 1 hour, 1.5 hours, 2 hours, 4 hours, 6hours & 24 hours.
Response Evaluation Criteria in Solid Tumours (RECIST) to explore the anti-tumour activity of NUC-3373 | Tumour assessment (CT scan/MRI scan) will be performed throughout study completion, every 8 weeks, an average of 6 per year.
  To explore the anti-tumour activity of NUC-3373 using Response Evaluation Criteria in Solid Tumours (RECIST) criteria in combination with tumour specific evaluation criteria which incorporates the relevant tumour markers (e.g. GCIG criteria utilising the Cancer Antigen 125 (CA125))

OTHER OUTCOMES:
Tertiary/Exploratory Objectives: Translational study to establish the expression of certain biomarkers in PBMCs and biopsy samples which may help to predict patients more likely to benefit from NUC-3373 over 5-FU. | through study completion, an average of 1 per year
  Potential biomarkers including but not limited to: Thymidine Phosphorylase (TP); Thymidine Kinase (TK); Thymidylate Synthase (TS); Dihydropyrimidine Dehydrogenase (DPD); Orotate Phosphoribosyl Transferase (OPRT); Cytidine Deaminase (CDA) and nucleoside / nucleobase transporters (hENT1, UraA). RNA will be analysed using a RNA scope
Tertiary/Exploratory Outcomes. To collect and bank samples for use in future ethically approved studies to explore potential stratification based on mutations e.g. KRas, VEGF and BRAF. RNA will be analysed using a RNA scope. | Screening/Baseline
  Where available, original diagnostic block will be recalled or patient can optionally consent for a biopsy to be performed prior to commencing study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah P Blagden, PhD, FRCP, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Belfast City Hospital, Belfast
  - Beatson, West of Scotland Cancer Centre, Glasgow
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spiliopoulou P, Kazmi F, Aroldi F, Holmes T, Thompson D, Griffiths L, Qi C, Parkes M, Lord S, Veal GJ, Harrison DJ, Coyle VM, Graham J, Jeffry Evans TR, Blagden SP. A phase I open-label, dose-escalation study of NUC-3373, a targeted thymidylate synthase inhibitor, in patients with advanced cancer (NuTide:301). J Exp Clin Cancer Res. 2024 Apr 2;43(1):100. doi: 10.1186/s13046-024-03010-1. PMID 38566164